CLINICAL TRIAL: NCT07378215
Title: The Effect of Corticosteroids on Quality of Life Following Total Hip Arthroplasty: HIPSTER Study
Acronym: HIPSTER
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Z-2025125; 2025-524368-39-00 (EU CTIS Number)
Record Dates: First submitted 2026-01-22; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Quality of Recovery; Health-Related Quality-of-Life; Quality of Life
Keywords: Hip Arthroplasty; Older adult patients; Dexamethasone; Enhanced Recovery After Surgery (ERAS); Quality of recovery; Quality of life
MeSH Terms: interventions — Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group 1 (Active Comparator): A single intraoperative dose of intravenous dexamethasone 5 mg
  Interventions: Drug: Dexamethasone (IV)
- Intervention group 2 (Active Comparator): A single intraoperative dose of intravenous dexamethasone 25 mg
  Interventions: Drug: Dexamethasone (IV)

INTERVENTIONS:
Drug: Dexamethasone (IV) — Dexamethasone 5 mg IV
  Other Names: Aacidexam (IV)
  Arms: Intervention group 1
Drug: Dexamethasone (IV) — Dexamethasone 25 mg IV
  Other Names: Aacidexam (IV)
  Arms: Intervention group 2

SUMMARY:
Total hip arthroplasty (THA) is a highly effective and commonly performed procedure for end-stage osteoarthritis. Perioperative inflammation contributes to postoperative pain, fatigue, and delayed recovery. Dexamethasone, a potent glucocorticoid with strong anti-inflammatory properties, is widely used in orthopedic surgery and incorporated into Enhanced Recovery After Surgery (ERAS) protocols for THA to reduce pain, PONV, and fatigue. While intermediate doses of dexamethasone (25 mg) are considered safe and beneficial in the short term, their long-term effects on health-related quality of life and persistent pain remain unclear.

Therefore, the main objective of the HIPSTER trial is to evaluate the effect of different doses of a single intraoperative intravenous dose of dexamethasone (5 mg versus 25 mg) on health-related quality of life up to three months after surgery.

DETAILED DESCRIPTION:
Total hip arthroplasty (THA) is a successful and cost-effective treatment for end-stage osteoarthritis and other degenerative hip conditions. It is one of the most frequently performed surgical procedures worldwide and continues to increase in volume each year, largely due to the growing population of older adults. Despite its effectiveness, THA is associated with significant surgical trauma that induces a pronounced inflammatory response, leading to postoperative pain, fatigue, postoperative nausea and vomiting (PONV), prolonged hospital stays, and delayed functional recovery. Prevention of postoperative inflammation can be a crucial cornerstone to optimize recovery and enhance outcomes after THA.

Dexamethasone, a potent and long-acting glucocorticoid with strong anti-inflammatory properties, is widely used in orthopedic surgery. It suppresses prostaglandin synthesis by downregulating cyclooxygenase-2 expression, thereby inhibiting cell adhesion factor expression and cytokine gene transcription. Dexamethasone also reduces neutrophil and macrophage exudation and activity at inflammatory sites, decreasing cellular adhesion and aggregation along vascular endothelium. Although dexamethasone has a short half-life of approximately 36-72 hours, by modulating the surgical stress response and its multiple downstream effects on inflammation, acute pain, nausea, and fatigue, it may also influence longer-term outcomes. Due to these mechanisms, dexamethasone has become an integral component of perioperative management in various surgical disciplines, including THA.

Previous studies have demonstrated that perioperative dexamethasone administration can attenuate inflammatory responses, reduce PONV, and acute postoperative pain and fatigue in patients undergoing THA. These short-term benefits translate into improved early postoperative recovery, which can be quantified using validated instruments such as the Quality of Recovery-15 (QoR-15) score. Consequently, dexamethasone is now commonly incorporated into Enhanced Recovery After Surgery (ERAS) protocols for THA. Intermediate glucocorticoid doses - equivalent to 25 mg of dexamethasone - are generally considered safe and are part of the standard of care in many arthroplasty centers performing primary THA.

While the short-term benefits of dexamethasone on postoperative inflammation, acute pain control, PONV reduction, early recovery, and hospital length of stay are well established in THA, concerns remain regarding its long-term safety profile. Several studies have reported potential adverse effects associated with intermediate to high doses, such as impaired sleep quality, immunosuppression, and possible wound-healing complications. Although glucocorticoids at the implemented doses have demonstrated efficacy in reducing acute postoperative pain, their role in preventing chronic postsurgical pain (CPSP) remains unclear, with some studies suggesting even a trend to persistent wound pain with higher doses of dexamethasone. Furthermore, the long-term effects of perioperative dexamethasone on health-related quality of life (HRQoL) following THA have not yet been systematically investigated.

As health-related quality of life, assessed by EQ-5D, is an important patient-reported outcome following anaesthesia and surgery, as emphasised in the StEP-COMPAC initiative, the effect of different doses of dexamethasone on health-related quality of life needs further investigation.

Therefore, the main objective of the HIPSTER trial is to evaluate the effect of different doses of a single intraoperative intravenous dose of dexamethasone (5 mg versus 25 mg) on health-related quality of life up to three months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* aged 60 years or older;
* scheduled for elective total hip arthroplasty;
* procedure under spinal anaesthesia.

Exclusion Criteria:

* hip revision surgery (reoperation);
* bilateral total hip arthroplasty during the same procedure;
* known hypersensitivity to dexamethasone or other corticosteroids;
* chronic systemic use of corticosteroids, defined as daily corticosteroid therapy for > 4 weeks within the last 3 months, with anticipated need for a perioperative stress dose of corticosteroids;
* active gastric of intestinal ulcers;
* lack of informed consent or inability to give informed consent;
* urgent, non-elective surgery.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Health-related quality of life (EQ5D5L) | Preoperative and postoperative day 30, day 60 and day 90
  The EQ5D is used for measuring health-related quality of life. EQ5D5L provides a single index value for health status which can be used to assess overall health. The descriptive profile consists of five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels of severity: no problems, slight problems, moderate problems, severe problems, or not able. Respondents select the level that best describes their current health status. The questionnaire will be taken preoperatively, on day 30, day 60 and day 90 following surgery.

SECONDARY OUTCOMES:
Quality of Recovery (QoR) | Preoperative and postoperative day 1, day 3 and day 5
  Quality of Recovery Score (QoR-15) is a patient-reported outcome measurement which will be used to assess the early postoperative health status of the patient after surgery and anesthesia, i.e. the quality of recovery. The score is arbitrary and ranges from 0 to 150, the higher the score the better the quality of recovery. QoR-15 will be assessed preoperatively and on day 1, day 3 and day 5 following surgery.
Health-related quality of life (EQ-VAS) | Preoperative and postoperative day 30, day 60 and day 90
  The EQ5D visual analog scale (VAS) EQ-VAS is used for measuring health-related quality of life. In the EQ-VAS respondents rate their current health status on a scale from 0 to 100, with 0 being the worst imaginable health and 100 being the best imaginable health state. The score will be taken preoperatively, on day 30, day 60 and day 90 following surgery.
Oxford Hip Score (OHS) | Postoperative day 30, day 60 and day 90
  The OHS is a joint-specific, patient-reported outcome measure designed to assess disability in patients undergoing total hip replacement surgery. It is a short 12-item survey where patients are asked to reflect on their pain and functional ability over the previous four weeks. There are two domains, pain and function, with six items in each. Each item has five possible responses. Item scores are summed to give a total score between 0 and 48. The lower the score, the better the outcome. The questionnaire will be done on day 30, day 60 and day 90 following surgery.
Brief Pain Inventory (BPI) | Preoperative and postoperative day 30, day 60 and day 90
  The BPI consists of 15 items and measures pain intensity and interference. The questionnaire comprises items regarding medications and analgesics, pain interference and intensity, relationships, mood, quality of life, and physical activities such as sleep, general activity and walking. Higher scores indicate greater severity and pain interference. The questionnaire will be done preoperative, on postoperative day 30, day 60 and day 90.
Chalder fatigue questionnaire (CFQ) | Preoperative and postoperative day 30, day 60 and day 90
  To assess general fatigue a fatigue questionnaire, the CFQ, will be taken preoperative and on day 30, day 60 and day 90 following surgery. The CFQ consists of 11 items that assess both physical and mental aspects of fatigue. Respondents rate each item ranging from 0 to 3, the scores are then totaled to provide a measure of overall fatigue, a higher score meaning more severe fatigue.

OTHER OUTCOMES:
NRS pain score at rest | Postoperative at 8 a.m. and 6 p.m. each day up to day 5 following surgery
  Numeric rating scale (NRS) pain score ranging from 0 to 10 with 0 reflecting no pain and 10 reflecting the worst pain at rest will be assessed postoperative at 8 a.m. and 6 p.m. each day up to day 5 following surgery.
NRS pain score at movement | Postoperative at 8 a.m. and 6 p.m. each day up to day 5 following surgery
  Numeric rating scale (NRS) pain score ranging from 0 to 10 with 0 reflecting no pain and 10 reflecting the worst pain at movement will be assessed postoperative at 8 a.m. and 6 p.m. each day up to day 5 following surgery.
NRS worst pain past 24 hours | Postoperative at 6 p.m. each day up to day 5 following surgery
  Numeric rating scale (NRS) pain score ranging from 0 to 10 with 0 reflecting no pain and 10 reflecting the worst pain in the past 24 hours will be assessed postoperative at 6 p.m. each day up to day 5 following surgery.
Use of analgesics in the past 24 hours | Postoperative at 6 p.m. each day up to day 5 following surgery
  Use of analgesics in the past 24 hours will be assessed postoperative at 6 p.m. each day up to day 5 following surgery.
Muscle strength (upper extremity) | Preoperative and postoperative day 1
  Postoperative muscle strength (upper extremity) will be assessed comparing the handgrip strength of the dominant hand, measured on day 1 following surgery as compared to the preoperative value.

CONTACTS AND LOCATIONS:
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No